CLINICAL TRIAL: NCT00005976
Title: Phase I/II Trial of Pyrazoloacridine and Carboplatin in Patients With Recurrent Glioma
Brief Title: Pyrazoloacridine Plus Carboplatin in Treating Patients With Recurrent Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01850; NCCTG-987254; CDR0000067963 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2003-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Gliosarcoma | interventions — Carboplatin; NSC 366140

ARMS (3):
- Arm I (Experimental): Patients receive carboplatin IV over 30 minutes and pyrazoloacridine IV over 3 hours on day 1. Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.
  Cohorts of 3-6 patients receive escalating doses of carboplatin and pyrazoloacridine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: carboplatin; Drug: pyrazoloacridine
- Arm II (Experimental): Patients receive the same treatment as given in study 1. Dose escalation is performed as in study 1 to determine the MTD in patients not receiving concurrent anticonvulsants.
  Interventions: Drug: carboplatin; Drug: pyrazoloacridine
- Arm III (Experimental): Patients receive the same treatment as given in studies 1 and 2 without dose escalation.
  Interventions: Drug: carboplatin; Drug: pyrazoloacridine

INTERVENTIONS:
Drug: carboplatin
Drug: pyrazoloacridine

SUMMARY:
Phase I/II trial to study the effectiveness of pyrazoloacridine plus carboplatin in treating patients who have recurrent glioma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of pyrazoloacridine plus carboplatin in patients with recurrent glioma.

II. Determine the toxic effects of this treatment regimen in these patients. III. Determine the safety of this treatment regimen at the recommended phase II dose in patients not receiving anticonvulsants.

IV. Determine the efficacy of this treatment regimen in these patients. V. Assess the pharmacokinetics and metabolism of pyrazoloacridine in these patients.

VI. Assess the response rate, time to progression, and time to death in patients treated with this regimen.

OUTLINE: This is a three-part, dose-escalation, multicenter study. Patients in study 3 are stratified according to concurrent anticonvulsants (yes vs no).

STUDY 1: (Study 1 closed as of 03/29/02) Patients receive carboplatin IV over 30 minutes and pyrazoloacridine IV over 3 hours on day 1. Treatment continues every 28 days in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of carboplatin and pyrazoloacridine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

STUDY 2: (Study 2 closed as of 03/29/02) Patients receive the same treatment as given in study 1. Dose escalation is performed as in study 1 to determine the MTD in patients not receiving concurrent anticonvulsants.

STUDY 3: Patients receive the same treatment as given in studies 1 and 2 without dose escalation.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually for 5 years.

PROJECTED ACCRUAL:

Study 1: A total of 3-21 patients will be accrued for this study within 6-20 months.

Study 2: A total of 3-12 patients will be accrued for this study within 3-18 months.

Study 3: A total of 12-37 patients will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary brain glioma

  * Diffuse astrocytoma
  * Gliosarcoma
  * Oligodendroglioma
  * Oligoastrocytoma
* Progressive disease after radiotherapy
* Measurable or evaluable disease by MRI or CT

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No congestive heart failure requiring therapy

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other active malignancy
* No other concurrent severe disease

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No more than 1 prior adjuvant chemotherapy regimen
* No prior polifeprosan 20 with carmustine implant (Gliadel wafer)
* Study 3 only:

  * 1 prior chemotherapy regimen for recurrent disease allowed
  * Prior nonplatinum-containing adjuvant chemotherapy allowed
  * Prior platinum-containing adjuvant chemotherapy allowed if disease progressed at least 6 months after last treatment

Endocrine therapy:

* Non-increasing dose of corticosteroids for at least 1 week allowed

Radiotherapy:

* At least 12 weeks since prior radiotherapy
* No prior stereotactic radiosurgery or interstitial brachytherapy unless at least one lesion outside of irradiated area

Surgery:

* No surgical resection since prior radiotherapy or chemotherapy unless evidence of disease progression or lesion outside of treatment site

Other:

* Study 1 only: (Study 1 closed as of 03/29/02)

  * Must be on anticonvulsants that can induce cytochrome P-450 (phenytoin, carbamazepine, barbiturates, or primidone)
* Study 2 only: (Study 2 closed as of 03/29/02)

  * No concurrent anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2000-05; Primary Completion 2006-12 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, MD, Study Chair — Mayo Clinic
Locations (23):
- United States (22):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Health Plaza, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Allan Blair Cancer Centre, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Galanis E, Buckner JC, Maurer MJ, Reid JM, Kuffel MJ, Ames MM, Scheithauer BW, Hammack JE, Pipoly G, Kuross SA. Phase I/II trial of pyrazoloacridine and carboplatin in patients with recurrent glioma: a North Central Cancer Treatment Group trial. Invest New Drugs. 2005 Oct;23(5):495-503. doi: 10.1007/s10637-005-2910-4. PMID 16133802